CLINICAL TRIAL: NCT03181750
Title: Apoyo Con Carino: (Support With Caring) Improving Palliative Care Outcomes for Latinos With Advanced Medical Illness
Brief Title: Apoyo Con Carino: Patient Navigation for Palliative Care for Non-Cancer Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Kaiser Permanente (Other); Denver Health Medical Center (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 16-1270; R01NR016467 (NIH)
Record Dates: First submitted 2017-06-05; First posted 2017-06-09 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Palliative Care
Keywords: Palliative Care; Latino; Patient Navigation

STUDY DESIGN:
Intervention Model Description: Multi-site Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Principal Investigator and outcomes assessor blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients and caregivers randomized to this arm will receive a packet of educational materials in English or Spanish. These materials are written at 5-6th grade reading level. The materials focus on advance care planning, pain and symptom management, and hospice care.
- Patient Navigator Intervention Group (Experimental): Patient and caregivers randomized to this arm will receive the same packet of educational materials. They will also receive at least 5 visits from a bicultural bilingual patient navigator. The navigator will utilize a annualized visit guide manual to lead discussions on advance care planning, pain and symptom management, and hospice care.
  Interventions: Behavioral: Patient Navigator Intervention Group

INTERVENTIONS:
Behavioral: Patient Navigator Intervention Group — Bicultural, bilingual navigators conducting home visits with patients and caregivers.
  Arms: Patient Navigator Intervention Group

SUMMARY:
Palliative care is a priority area of focus for the National Institute of Nursing Research. Despite the evidence-based benefits of palliative care, access remains limited, especially in poor urban and rural settings. Cultural and linguistic barriers may also increase disparities in palliative care for Latinos. Due to a nationwide shortage of palliative care providers and the unique cultural preferences and values of patients, our innovative study has the potential to improve palliative care outcomes and reduce health disparities in both urban and rural underserved communities.

DETAILED DESCRIPTION:
Latinos are more likely to experience uncontrolled pain, institutional death, and are less likely to engage in advance care planning. Efforts to increase access to palliative care must maximize primary palliative care and community based models to meet the ever growing need in a culturally-sensitive and congruent manner. Patient navigator interventions are community based, culturally tailored models of care and have been successfully implemented to improve disease prevention, early diagnosis and treatment. The investigators have developed and implemented a patient navigation intervention to improve palliative care outcomes for seriously ill hospitalized Latinos. They have demonstrated feasibility and early findings suggest this intervention can improve palliative care outcomes for Latinos with advanced cancer. Building on this prior research, the investigators propose a fully powered randomized controlled trial to determine the effectiveness of the manualized patient navigator intervention in a non-cancer population. A total of 240 Latino adults with non-cancer, advanced medical illness enrolled from 8 urban and 4 rural clinical sites will be randomized to the intervention group (5 palliative care-related patient navigator visits plus educational materials) or control group (usual care plus educational materials). Participants randomized to the intervention group will demonstrate better quality of life, will be more likely to have a palliative approach to their care, have higher rates of advance care planning, better pain and symptom control, and higher rates of hospice utilization compared to the control group). They will conduct a cost analysis of the patient navigator intervention by comparing direct costs of the intervention and cost and utilization of health care system resources across the study arms. Participants randomized to the intervention will have lower costs in the 6 months following study enrollment compared to participants in the control arm. Decedent participants randomized to the intervention will have lower costs in the last 3 months of life compared to decedent participants in the control arm. For the intervention visits, bicultural, bilingual navigators (guias) integrate core Latino values, while addressing barriers to a palliative approach through education, culturally tailored messaging, and patient activation. Patients will be interviewed at baseline and 3 months using the QUAL-E quality of life scale, Brief Pain Inventory, Edmonton Symptom Assessment Scale, and the Patient Navigator Process and Outcomes Measure. Medical records will be reviewed to assess advance directive completion, hospice and health care utilization and intensity of care at the end of life. This culturally tailored, evidence-based, theory driven, highly innovative patient navigation intervention has significant potential to improve palliative care for Latinos, and facilitate true health equity in palliative and end of life care.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Latino
* Age 18-90 years
* Not referred or enrolled in hospice care
* Meeting medium to high risk for death at 1 year using the CARING criteria (although excluding patients with cancer diagnosis)

OR

* If health care provider answers "no" to the question: "Would you be surprised if this patient died in the next year?"

Exclusion Criteria:

* Cancer diagnosis
* Referred or receiving hospice care
* Pregnant
* Incarcerated
* Lacking decisional capacity

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2017-06-02 (Actual); Primary Completion 2020-12-09 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
FACIT-Quality of Life Assessment | 3 months post enrollment
  Validated and responsive Quality of Life measure
Caregiver Reaction Assessment | 3 months post enrollment
  For caregivers: A validated measure of caregiver burden and positive meaning finding for caregivers

SECONDARY OUTCOMES:
Brief Pain Inventory | 3 months post enrollment
  A validated pain assessment measure
Edmonton Symptom Assessment Scale | 3 months post enrollment
  A validated symptom assessment scale
Patient Navigation Process and Outcome Measure | 3 months post enrollment
  A satisfaction and process measure developed for the patient navigator intervention
Advance Care Planning | 6 months post enrollment
  chart review to document presence of advance directive
Hospice Utilization | month 46 of the study
  hospice length of stay in days
Advance Care Planning Engagement Survey | 3 months post enrollment
  A validated measure of readiness to engage in advance care planning

OTHER OUTCOMES:
Cost Effectiveness of the Intervention | 6 months post intervention
  costs of providing the intervention versus costs of utilization of health care with and without intervention
Cost Effectiveness of the Intervention for End of Life | last 3 months of life
  costs of providing the intervention versus costs of utilization of health care with and without intervention for those patients who die during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Stacy M Fischer, MD, Principal Investigator — University of Colorado, Denver
Locations (6):
- United States (6):
  - University of Colorado Health Central, Aurora, Colorado
  - University of Colorado Health, Colorado Springs, Colorado
  - Centura Health, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente Colorado-N/S/W, Denver, Colorado
  - University of Colorado Health North, Fort Collins, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fischer SM, Min SJ, Kline DM, Lester K, Gozansky W, Schifeling C, Himberger J, Lopez J, Fink RM. Patient Navigator Intervention to Improve Palliative Care Outcomes for Hispanic Patients With Serious Noncancer Illness: A Randomized Clinical Trial. JAMA Intern Med. 2024 Apr 1;184(4):384-393. doi: 10.1001/jamainternmed.2023.8145. PMID 38345793
- [Derived] Fink RM, Valenti KG, Kline DM, Fischer SM. Reality of Family Caregiving for Hispanics With Alzheimer's Disease and Related Dementias: A Qualitative Analysis. J Palliat Med. 2023 Dec;26(12):1618-1626. doi: 10.1089/jpm.2023.0008. Epub 2023 Jun 13. PMID 37311202